CLINICAL TRIAL: NCT06575491
Title: Comparative Evaluation of Ultrasound Guided Supraclavicular and Infraclavicular Subclavian Venous Catheterization in Pediatric
Brief Title: Ultrasound Guided Supraclavicular and Infraclavicular Subclavian vs Catheterization in Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Radi Mohamed Radi Mostafa, Resident of Anesthesiology, Surgical Intensive Care, Faculty of Medicine, Al-Azhar University, Cairo, Egypt., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0377/2023
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Ultrasound Guided; Supraclavicular; Infraclavicular; Subclavian; Venous Catheterization; Pediatric

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular group (Experimental): Patients submitted to Supraclavicular approach for ultrasound-guided Subclavian veinous catheterization.
  Interventions: Device: Ultrasound-guided supraclavicular approach
- Infraclavicular group (Experimental): Patients submitted to Infraclavicular approach for ultrasound-guided Subclavian veinous catheterization.
  Interventions: Device: Ultrasound-guided infraclavicular approach

INTERVENTIONS:
Device: Ultrasound-guided supraclavicular approach — Patients submitted to Supraclavicular approach for ultrasound-guided Subclavian veinous catheterization.
  Arms: Supraclavicular group
Device: Ultrasound-guided infraclavicular approach — Patients submitted to Infraclavicular approach for ultrasound-guided Subclavian veinous catheterization.
  Arms: Infraclavicular group

SUMMARY:
The aim of this study was to compare between ultrasound-guided supraclavicular and infraclavicular approaches for subclavian venous catheterization in pediatric to get clinical practice of rapid, accurate central venous catheter, insertion and less Complications.

DETAILED DESCRIPTION:
Vascular access in children can be challenging. There is a considerable body of evidence supporting the use of ultrasound to aid central venous access in adults, but less so in children. Benefits for experienced operators may be small, but there is evidence of benefit for those acquiring skills and for less frequent operators.

Central venous catheter (CVC) placement is one of the most important invasive procedures in the intensive care for children of all ages. And health care outcomes largely depend on the success of its implementation. There are a large number of historically and clinically significant methods of central venous catheterization, and the advantages and disadvantages of each of them have been discussed for many years.

Ultrasonography is becoming an increasingly useful adjunct in the placement of Percutaneous central lines.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 4 to 12 years.
* Both sexes.
* All children who need central venous line insertion.
* Intra-operative Hemodynamic monitoring.
* Volume and Inotrope Resuscitation.
* Difficult Peripheral IV Access.
* Intravenous Nutrition and Medications.

Exclusion Criteria:

* Coagulopathy.
* Distorted anatomy.
* Infection systemic or cutaneous near the proposed Point of insertion.
* Skeletal deformity.
* History of previous neck surgery.
* Head and neck mass.
* Guardian Refusal.
* Pneumothorax Or Hemothorax.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Puncture time | Interoperatively
  Puncture time was recorded.

SECONDARY OUTCOMES:
Total access time | Interoperatively
  Total access time was recorded
First attempt success rate | Interoperatively
  First attempt success rate was recorded
Quality of needle visualization | Interoperatively
  Quality of needle visualization was recorded
Incidence of complication | 24 hours postoperatively
  Incidence of complication was recorded such as complication rates.failure rate haematoma, pneumothorax

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author.